CLINICAL TRIAL: NCT00457080
Title: Application of Capnography Monitoring on the General Care Nursing Unit
Acronym: ETCO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Health Resources (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CAPNO-P806
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-07

CONDITIONS: Postoperative Complications
Keywords: capnography; safety; opioids; respiratory depression; postoperative; orthopedic; OSA; apnea
MeSH Terms: conditions — Postoperative Complications; Respiratory Insufficiency; Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Alaris ETCO2 monitor - cont. resp. rate, & apnea events

SUMMARY:
The aim of this study is to increase the detection of undiagnosed obstructive sleep apnea (OSA) and secondly to increase the sensitivity for detection of respiratory depression (< 6 breaths per minute) in post operative patients on the general care nursing unit.

DETAILED DESCRIPTION:
Measures: This is an IRB approved prospective trial beginning with randomization in the post anesthesia care unit (PACU) and continuing for thirty six hours post orthopedic surgical procedure. The patients are randomized into a capnography or standard of care group and the percentage of newly identified OSA patients were measured in each group using the criteria set forth by 2006 American Society of Anesthesiologist practice guideline (Anesthesiology 2006; 104:1081-93).

Background/Changes: Hospital complications are three times higher in patients with obstructive sleep apnea and the majority of these complications are related to opioid induced respiratory depression (Mayo Clin Proc Sept 2001:897-905). American Society of Anesthesiologist 2006 practice guideline for perioperative management of patients with obstructive sleep apnea (Anesthesiology 2006; 104:1081-93) lists the criteria for identifying undiagnosed obstructive sleep apnea. One of the risk factors in the guideline lists apnea (pauses in breathing). Capnography measures apnea episodes and continuously monitors respiration rate.

As previously described, five percent of the general population has obstructive sleep apnea (OSA) and the prevalence among patients requiring surgery is 9% (NEJM 1993; 328:1230-1235). Between 50-80% of OSA individuals are undiagnosed when presenting for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Orthopedic surgical procedure
* Respiration rate < 10 breaths per minute requiring supplement oxygen
* One of the following:

  * body mass index >30
  * history of snoring
  * basal rate of opioid, and
  * one event of RR <10 in the post anesthesia care unit.

Exclusion Criteria:

* COPD
* < 18 y/o
* A diagnosis of obstructive sleep apnea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-10; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Increase the detection of undiagnosed obstructive sleep apnea (OSA)

SECONDARY OUTCOMES:
Increase the sensitivity for detection of respiratory depression (< 6 breaths per minute) in post operative patients on the general care nursing unit

CONTACTS AND LOCATIONS:
Overall Officials: Rob W Hutchison, Principal Investigator — Texas Health Resources
Locations (1):
- Presbyterian Hospital of Dallas, Dallas, Texas, United States

REFERENCES:
- [Background] Hutchison R. Capnography monitoring during opioid PCA administration. J Opioid Manag. 2006 Jul-Aug;2(4):207-8. doi: 10.5055/jom.2006.0032. No abstract available. PMID 17319481
- [Background] Kirk VG, Batuyong ED, Bohn SG. Transcutaneous carbon dioxide monitoring and capnography during pediatric polysomnography. Sleep. 2006 Dec;29(12):1601-8. doi: 10.1093/sleep/29.12.1601. PMID 17252891
- [Background] Krauss B, Hess DR. Capnography for procedural sedation and analgesia in the emergency department. Ann Emerg Med. 2007 Aug;50(2):172-81. doi: 10.1016/j.annemergmed.2006.10.016. Epub 2007 Jan 12. PMID 17222941
- [Background] Anderson JL, Junkins E, Pribble C, Guenther E. Capnography and depth of sedation during propofol sedation in children. Ann Emerg Med. 2007 Jan;49(1):9-13. doi: 10.1016/j.annemergmed.2006.06.011. Epub 2006 Aug 17. PMID 17141136
- [Background] Lightdale JR, Goldmann DA, Feldman HA, Newburg AR, DiNardo JA, Fox VL. Microstream capnography improves patient monitoring during moderate sedation: a randomized, controlled trial. Pediatrics. 2006 Jun;117(6):e1170-8. doi: 10.1542/peds.2005-1709. Epub 2006 May 15. PMID 16702250
- [Background] Anderson MR. Capnography: considerations for its use in the emergency department. J Emerg Nurs. 2006 Apr;32(2):149-53. doi: 10.1016/j.jen.2005.12.025. No abstract available. PMID 16580478
- [Background] Corbo J, Bijur P, Lahn M, Gallagher EJ. Concordance between capnography and arterial blood gas measurements of carbon dioxide in acute asthma. Ann Emerg Med. 2005 Oct;46(4):323-7. doi: 10.1016/j.annemergmed.2004.12.005. PMID 16187465
- [Background] Verschuren F, Heinonen E, Clause D, Zech F, Reynaert MS, Liistro G. Volumetric capnography: reliability and reproducibility in spontaneously breathing patients. Clin Physiol Funct Imaging. 2005 Sep;25(5):275-80. doi: 10.1111/j.1475-097X.2005.00620.x. PMID 16117730
- [Background] Fisher QA. Can capnography substitute for auscultation in sedation cases? Anesth Analg. 2005 May;100(5):1546. doi: 10.1213/01.ANE.0000151470.50760.4A. No abstract available. PMID 15845739
- [Background] Hatlestad D. Capnography in sedation and pain management. Emerg Med Serv. 2005 Mar;34(3):65-9. PMID 15839539
- [Background] Eisenbacher S, Heard L. Capnography in the gastroenterology lab. Gastroenterol Nurs. 2005 Mar-Apr;28(2):99-105; quiz 105-6. doi: 10.1097/00001610-200503000-00003. PMID 15832109
- [Background] Dziewas R, Hopmann B, Humpert M, Bontert M, Dittrich R, Ludemann P, Young P, Ringelstein EB, Nabavi DG. Capnography screening for sleep apnea in patients with acute stroke. Neurol Res. 2005 Jan;27(1):83-7. doi: 10.1179/016164105X18359. PMID 15829165
- [Background] Engoren M, Plewa M, O'Hara D, Kline JA. Evaluation of capnography using a genetic algorithm to predict PaCO2. Chest. 2005 Feb;127(2):579-84. doi: 10.1378/chest.127.2.579. PMID 15705999